CLINICAL TRIAL: NCT03368027
Title: Effectiveness of a Program for Coping With Psychological Stress on Stress, Psychopathology, Self-efficacy, Resilience, Social Support and Visual Field in People With Retinitis Pigmentosa
Brief Title: Effectiveness of a Cognitive-behavioral Program of Coping With Psychological Stress in People With Retinitis Pigmentosa
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Retinitis pigmentosa RCT
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Vision Disorders; Stress, Psychological; Psychopathy; Self Efficacy
Keywords: Vision Disorders; Stress, Psychological
MeSH Terms: conditions — Vision Disorders; Stress, Psychological; Antisocial Personality Disorder | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress management program (Experimental): A cognitive-behavioral program of coping with psychological stress for 3 months (with a total of 12 sessions), one session per week, with a duration of 90 minutes per session.
  Interventions: Behavioral: A cognitive-behavioral intervention program
- Standard intervention (Active Comparator): Usual activities performed in the association where they attend (supervised by a psychologist) for 3 months (with a total of 12 sessions), one session per week, with a duration of 90 minutes per session.
  Interventions: Other: Standard intervention

INTERVENTIONS:
Behavioral: A cognitive-behavioral intervention program — In this program, participants receive a training of assertive skills, social skills, acceptance, among other psychological aspects.
  Other Names: Cognitive-behavioral program
  Arms: Stress management program
Other: Standard intervention — Participants receive different activities conducted by a psychologist in the association where the attend.
  Other Names: Control group
  Arms: Standard intervention

SUMMARY:
The aim of this study is to evaluate the efficacy of cognitive - behavioral therapy for the control of psychopathological stress and the disease of people with Retinitis Pigmentosa (RP).

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the efficacy of cognitive - behavioral therapy for the control of psychopathological stress and the disease of people with Retinitis Pigmentosa (RP) on aspects such as vulnerability to stress, perceived stress, psychopathological state, general self-efficacy, resilience, satisfaction with social support and visual field. This study has two groups: 1) cognitive - behavioral therapy group, and 2) Standard intervention or control group. The two interventions will be conducted for 3 months (with a total of 12 sessions), one session per week, with a duration of 90 minutes per session.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Retinitis Pigmentosa (legally blind RP patients).
* meet the membership criteria of the Spanish National Association of ONCE.
* having a reduction of the visual field of at least 10 degrees in both eyes
* having an age between 18 and 65 years.

Exclusion Criteria:

* no visual remainders (advanced retinosis).
* no studies.
* cognitive impairment, determined by the Spanish Mini-Mental State Examination - MMSE test.
* mobility problems
* high risk of falls associated with retinosis, measured by the Morse scale, with a score over 50 points.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in vulnerability to stress at 12 weeks | Twelve weeks
  This scale registeres the aspects that influence the ability to deal with stress

SECONDARY OUTCOMES:
Change from Baseline in Perceived stress scale at 12 weeks | Twelve weeks
  This scale evaluates the degree to which situations in one's life are appraised as stressful
Change from Baseline in Symptom Checklist-90-Revised Questionnaire at 12 weeks | Twelve weeks
  This instrument is a 90-item self-report symptom inventory developed by Leonard R. Derogatis in the mid-1970s to measure psychological symptoms and psychological distress.
Change from Baseline in General Self efficacy scale at 12 weeks | Twelve weeks
  This scale assesses people's stable believe about their ability to appropriately manage a wide kind of life stressors
Change from Baseline in Connor-Davidson Resilience Scale at 12 weeks | Twelve weeks
  This scale evaluates stress coping ability.
Change from Baseline in Social support questionnaire at 12 weeks | Twelve weeks
  This instrument evaluates perceived Social support.
Change from Baseline in Visual Field Test at 12 weeks | Twelve weeks
  This method evaluates the visual field of two eyes

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Pérez Mármol, PhD, Principal Investigator — Department of Physiotherapy. Faculty of Health Sciences, University of Granada
Locations (1):
- José Manuel Pérez Mármol, Granada, Spain

IPD SHARING:
Plan to Share IPD: No